CLINICAL TRIAL: NCT06454396
Title: A Real-world Clinical Study Based on a Decentralized Arteriovenous Endovascular Fistula Data System - Effectiveness and Health Economics of Endoluminal Treatment of Autologous Arteriovenous Endovascular Fistula Failure
Brief Title: Effectiveness and Health Economics of Endoluminal Treatment of Autologous Arteriovenous Endovascular Fistula Failure
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: The AVF study
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Hemodialysis Access Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Endovascular therapy — Endovascular therapy is a minimally invasive interventional approach that utilizes the vascular system as a pathway to access and treat various pathological conditions within the body. By employing specialized catheters and devices, endovascular techniques enable precise delivery of therapeutic agents or interventional procedures directly to the target site, without the need for conventional open surgery.

SUMMARY:
This study was aimed at evaluating the efficacy of different endovascular treatments for early and mid-stage clinical interventions in patients with autologous arteriovenous fistulae loss of function and the corresponding health economic value.

DETAILED DESCRIPTION:
This is a prospective, single-center, real-world study intended to understand the clinical intervention efficacy and health economic value of various real-world endovascular treatments for autologous arteriovenous endovascular fistulae failure in a target lesion defined as the hemodialysis access inflow tract (arterial, anastomotic, and inflection), intermediate segment, and outflow tract vein. The study will enroll 480 patients with autologous arteriovenous endovascular fistulae that have failed during the period 2023/1-2024/12, in a single center. They will be divided into subgroups according to different treatment modalities, such as balloon dilatation alone group, medicated balloon group, and stent implantation group. The main observations were the technical success rate of various endoluminal treatment methods, perioperative major adverse events, and symptom-driven target lesion re-intervention rate, target vessel patency rate, and total hospitalization expenditures related to the target lesion at 1, 6, 12, 18, and 24 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis patients over 18 years of age and under 80 years of age
2. Autologous arteriovenous fistula cannot be used in patients completing haemodialysis
3. The guidewire must pass through at least the stenosis of the endovascular fistula on the side of the lesion and undergo further endovascular treatment before enrolment, and this study does not limit the form of the guidewire passing through the target lesion.
4. Patients who have failed to open the initial target lesion and are successful on a second attempt at endoluminal therapy may still be enrolled.
5. Subjects and their legal representatives are able to understand the purpose of the study, participate voluntarily and sign an informed consent form, and are willing to be followed up at specific points in time.

Exclusion Criteria:

1. Planned kidney transplant or conversion to peritoneal dialysis
2. Women who are pregnant, breastfeeding or planning to become pregnant during the study period
3. Recent (within 30 days) or planned surgical procedure for haemodialysis access
4. Allergy or contraindication to heparin, contrast media, antiplatelet drugs
5. Patients who have participated in a clinical trial of a drug or other medical device that interferes with this clinical trial within the last 3 months.
6. Patients with a history of coagulation disorders or other haematological disorders
7. Patients with other conditions that may make the trial difficult or significantly shorten the patient's life expectancy (<2 years), e.g. tumours, severe liver disease, cardiac insufficiency, etc., or patients with a life expectancy of less than 6 months.
8. Patients unable or unwilling to participate in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dysfunctional autogenous arteriovenous fistula patient:
  A stenosis in a hemodialysis access with significant hemodynamic changes: Based on angiography/ultrasound evaluation, the target lesion stenosis is ≥50%, and is accompanied by one or more of the following clinical and physiological abnormalities: natural fistula blood flow <480ml/min; unable to meet the required blood flow for the dialysis prescription; thrombosis in the autogenous arteriovenous fistula; elevated venous pressure during dialysis; difficult cannulation; decreased dialysis adequacy; and abnormal signs in the fistula, etc.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically-driven target lesion re-intervention | 1-month；6-month；12-month；18-month；24-month
  Clinically-driven target lesion re-intervention refers to a repeat procedure performed on a previously treated lesion due to the recurrence of symptoms or other clinical indications, rather than being routinely scheduled.

SECONDARY OUTCOMES:
target lesion primary patency | 1-month；6-month；12-month；18-month；24-month
  Target lesion primary patency refers to the treated lesion site remaining open and unobstructed without the need for any additional revascularization procedure during the follow-up period.
target lesion assisted primary patency | 1-month；6-month；12-month；18-month；24-month
  Target lesion assisted primary patency refers to the treated lesion site remaining patent (open) during the follow-up period, but requiring an additional revascularization procedure, such as percutaneous transluminal angioplasty, to maintain patency of the target lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided